CLINICAL TRIAL: NCT06901674
Title: Stimulating the Cochlear Apex Without Longer Electrodes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-01964; 5R21DC019743-02 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Deafness With a Cochlear Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Apical ground electrode (Experimental): Participants in this group will have already received a cochlear implant using the new approach or be receiving a cochlear implant with the new approach.
  Interventions: Procedure: Modified surgical approach; Device: Cochlear Nucleus CI632 cochlear implant
- Standard location ground electrode (Active Comparator): Participants in this group have received a cochlear implant with the typical ground electrode placement.
  Interventions: Device: Cochlear Nucleus CI632 cochlear implant

INTERVENTIONS:
Procedure: Modified surgical approach — An electrode typically placed under the temporalis muscle will be placed into the cochlear helicotrema instead.
  Arms: Apical ground electrode
Device: Cochlear Nucleus CI632 cochlear implant — Cochlear implant (CI) system where stimulation from one of the intracochear electrodes is grounded via one of two (or both) extra cochlear electrodes in the device.

SUMMARY:
The most common cochlear implant intervention provides an electrode array that stimulates less than half of the length of the cochlea, leaving the regions which represent lower frequencies in the normally functioning ear unstimulated. Providing stimulation over the entire cochlea has the potential to improve speech understanding, sound quality, as well as spectral and temporal representation. Increasing the length of the electrode array to cover a greater portion of the cochlea has many potential issues, including increased damage to the cochlea and probability of incomplete insertions. In this study, a new technique is being investigated that allows stimulation across the entire cochlear extent without increasing the length of the electrode array. The purpose of this study is to evaluate the benefit of the new technique on speech understanding outcomes. Additionally, the study will investigate the new configuration to explore how the auditory system encodes temporal and spectral information.

ELIGIBILITY:
Inclusion Criteria:

* Participants in this study must have already been evaluated at the NYU cochlear implant center as being eligible for a cochlear implant.
* They must have decided to receive a cochlear implant manufactured by Cochlear Limited and have been diagnosed with a moderate to profound sensorineural hearing loss in the ear to be implanted.
* Individuals who have already been implanted with a cochlear implant manufactured by Cochlear Limited with or without this new approach may also participate in this study.

Exclusion Criteria:

* They are under the age of 18
* They have not been diagnosed with a moderate to profound sensorineural hearing loss in the ear to be implanted
* Have >15 years of profound deafness
* Have not chosen to receive a cochlear implant manufactured by Cochlear Limited
* Are pregnant or plan to conceive within 6 months of consenting

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Upper Limit of Rate Pitch Perception for Cochlear Implant Stimuli | Month 12
  The upper limit of rate pitch perception will be evaluated for Apex-monopolar (MP), 22-Apex, 22-MP, and 11-MP cochlear implant stimuli using a 3-up 1-down 2-interval forced-choice adaptive task. The task measures the highest modulation frequency perceived as a lower pitch compared to a rate 5 semitones higher. A series of 750-ms, 5000-pps pulse trains with 100% amplitude modulation will be presented at a loudness-balanced most-comfortable level. The upper limit will be estimated from the average modulation frequency of the last 6 reversals across 10 trials per stimulation site.
Mean pitch rank | Month 12
  Pitch-ranking will be done using a 2-interval forced-choice protocol in which the pitch of a newly selected stimulus is ranked relative to the stimulus in the middle of a pitch-rank order list. Depending on the ranked pitch direction, this stimulus is repositioned in the pitch-rank order list and ranked against a neighboring stimulus until the correct position in the list is determined. This process repeated until all stimuli are successfully pitch ranked. A complete set of pitch ranks are measured 10 times allowing for the calculation of a mean rank and 95% confidence interval for the rank of each interval.
Percentage of Consonant-Nucleus-Consonant (CNC) words correctly repeated | Month 12
  Speech perception will be assessed using CNC word lists, a common method for evaluating monosyllabic word recognition. The CNC Monosyllabic Word Test includes 10 lists of 50 words. The word test score range typically used is between 10% and 60% correct in the ear to be implanted, and equal to or better than that ear in the contralateral ear, but not better than 80% correct.

CONTACTS AND LOCATIONS:
Overall Officials: David M. Landsberger, Ph.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to:David.landsberger@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to David.landsberger@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.